CLINICAL TRIAL: NCT02541526
Title: Mirtazapine as a Treatment for Co-Occurring Opioid and Amphetamine Type Stimulant Dependence (COATS) in Malaysia
Brief Title: Mirtazapine as a Treatment for Co-Occurring Opioid and ATS Dependence in Malaysia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Vicknasingam B Kasinather, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00004494b
Record Dates: First submitted 2015-06-29; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Heroin Dependence; Amphetamine Dependence
Keywords: amphetamine type stimulant dependence; mirtazepine
MeSH Terms: conditions — Heroin Dependence; Amphetamine-Related Disorders | interventions — Mirtazapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mirtazapine (Experimental): 30 mg mirtazepine will be given to patients on day 6 of their treatment for a period pf 3 days to observe for tolerability followed by 60 mg from day 9 of treatment until the end of the study (16 weeks).
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): matched placebo mirtazapine capsules will be given to patients in this group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — One capsule (15 mg) oral mirtazepine daily will be started on day six of treatment for a period of 3 days followed by two capsules (30 mg) daily for a period of four months
  Other Names: Remeron
  Arms: mirtazapine
Drug: Placebo — Similar capsule containing placebo will be started on day six of treatment for a period of 3 days followed by two capsules of placebo daily for a period of four months
  Other Names: Sugar
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate tolerability, acceptability and potential efficacy of 4 months of maintenance treatment with Mirtazapine as compared to placebo for patients with co-occurring amphetamine-type stimulant and opioid dependence (COATS) receiving buprenorphine maintenance treatment (BMT) in Kota Bharu.

DETAILED DESCRIPTION:
Amphetamine type stimulant (ATS) and opioid abuse, dependence and injection drug use (IDU) are major public health problem in Malaysia and nearby countries (including China, Indonesia, Thailand, Vietnam, Myamar, and Cambodia) and are the major drivers of the HIV/AIDS epidemic in these countries.1 Opioids (predominantly heroin, morphine, or, to a lesser extent, opium) are the primary drugs of abuse for most drug users in Malaysia and the region. There are more than 300,000 registered drug users in Malaysia (estimated >500,000 total); most are opioid dependent and current IDUs; 25-30% of IDUs are infected with HIV; and IDU accounts for 70% of HIV infections in Malaysia (91,360 registered HIV+ between 1986 and 2010).6 Over the past decade, ATS has also emerged as an additional major drug problem. Globally, ATS is now the second most commonly used illicit drug type (after marijuana) and is more widely used than heroin.1-6, 2 ATS abuse is especially prevalent and problematic in the Asian region, where ATS production, use, drug seizures, demand for treatment, and medical consequences have continued to increase through the most recent 2011 report. Laboratories producing ATS have been identified in more than half of the countries in the region; large scale laboratories capable of industrial-scale manufacture have been found in Malaysia, China, and Indonesia. Injection of methamphetamine has been reported in Malaysia, Indonesia, Thailand, and Singapore. Data from our recently completed studies and others document a rapid rise in the prevalence of ATS use among opioid IDUs over the past decade; in the most recent survey of out-of-treatment heroin IDUs in cities across Malaysia, more than 60% report current ATS use, and 29% inject ATS.

ATS use is associated with increased behavioral risks of HIV transmission (even in already at high risk opioid IDUs), In our earlier studies conducted in Malaysia, we found an increased prevalence of HIV, increased needle sharing and risky sexual behaviors among opiate dependent IDUs who also reported lifetime use, as compared to opioid IDUs who do not use ATS. ATS use is also associated with poor anti-retroviral medication adherence. ATS use exacerbates HIV transmission risk through a number of mechanisms: ATS users report engaging in more frequent and more risky sexual behaviors while using ATS3, and in more frequent IDU and equipment sharing. ATS use may enhance sexual desire, an effect many opiate dependent individuals (or individuals maintained on MMT) may particularly desire because of opioid-induced hypogonadism and a resulting loss of libido. ATS is also associated with impairments of mood and executive functioning that may persist for prolonged periods and may contribute to relapse to drug use, IDU, and other high risk behaviors. Consequently, it is critical to develop and evaluate treatments to reduce opioid and ATS use, IDU, and HIV transmission risk among individuals with COATS.

Located in the northeastern region of peninsular Malaysia, bordering Thailand, Kota Bharu, the densely populated and fast growing capital city of Kelantan state and site of the proposed study, provides a unique opportunity for conducting the proposed study. Kota Bharu and Kelantan are experiencing the most severe problems with illicit opioid and ATS use, IDU and HIV in Malaysia. The number of individuals arrested annually for ATS in Kelantan increased over the past 5 years from 2900 in 2007 to 5300 in 2010. For the past 5 years, Kelantan has also led Malaysia in having the highest population prevalence of HIV infection (47 per 100,000 in 2008, nearly 4 times the prevalence reported for the rest of Malaysia). Kelantan also has the highest number of women with HIV in Malaysia (more than 1200 reported in 2008), suggesting that HIV is making the transition to the general population. A large proportion of treatment seeking drug users in Kelantan are HIV + and are susceptible to high mortality: Since MMT was first introduced in Kelantan in 2006, 623 of 1128 (53%) MMT patients with known HIV status were HIV+, and 126 of 1148 patients enrolled in MMT died following enrollment [Personal communication, Dr. Hazura BT Mat Zubir, Kelantan Health Department, December 5, 2011].

Currently, there are no proven efficacious medications for treating Amphetamine type stimulants (ATS) dependence or co-occurring opioid and ATS dependence (COATS). Although opioid agonist maintenance treatment (OMT) with methadone and buprenorphine are efficacious for treating opioid dependence and reducing HIV transmission risk, many patients continue opioid and ATS use and HIV risk behaviors during OMT, and the overall good efficacy of OMT is substantially reduced for patients with COATS. Patients with COATS are also at particularly high risk for HIV infection or transmission due to both drug- and sex-related behaviours.

Pharmacology of Mirtazapine

Mirtazapine is a novel antidepressant agent that acts as an antagonist of inhibitory alpha 2 adrenergic presynaptic receptors and alpha 2 heteroreceptors in the serotenergic nerve terminals. Mirtazapine increase norepinephrine release and selective serotonergic (5-HT1A) transmission by acting as antagonist at alpha 2 adrenergic presynaptic receptor which resulted in increase of norepinephrine release and acting on alpha 2 heteroreceptors in the serotonergic nerve terminals which increase serotonin release. Mirtazapine selectively act on 5-HT1A neurotransmission by blocking on 5-HT2 and 5-HT3 receptors. It also enhances frontocortical release dopaminergic transmission via 5-HT1A activation and dopamine release in the prefrontal cortex via blockage of alpha 2 adrenergic and 5HT2C receptors.

Mirtazapine was initially evaluated as a potential treatment for ATS withdrawal based on its pharmacological effect on norepinephrine, serotonin and dopamine neurotransmissions which has been effectively shown to treat sleep problems, anxiety and depression. Recent studies in human and animal evidenced that mirtazapine has a promising role for the treating ATS dependence. Two small pilot 2,4 showed that mirtazapine improved sleep and reduced ATS withdrawal symptoms. Another study 5 showed that mirtazapine was not as effective as Modafinil in improving sleep or ATS withdrawal symptoms. Preclinical studies in animals provide additional support for the potential efficacy of mirtazapine in treating ATS dependence. Cue elicited drug craving is an important mechanism underlying relapse following abstinence and its modulation in brain involved the limbic reward region and mediated by both glutaminergic and dopaminergic neurotransmission. Studies in animal models showed that mirtazapine block cue elicited behavioural response which is believed due to the modulation effect of mirtazapine on noradrenergic and serotonergis systems. Repeated mirtazapine treatment eliminates ATS-induced conditioned place preference in rats suggesting that it may disrupt ATS associated memory consolidation or reconsolidation following re exposure.

Mirtazapine is one of the most promising medication for the treatment ATS dependence and it's preliminary efficacy has been shown in a double blind, randomized, placebo controlled clinical trial. The study conducted with 60 actively using , ATS dependent men who have sex with men (MSM), found that the addition of mirtazapine to substance abuse counselling decreased ATS use and sexual risk behaviours. Mirtazapine is a safe drug that has no serious adverse effect. Potential adverse effects of Mirtazapine include decreased appetite, weight loss, insomnia, nausea and vomiting, diarrhoea, urinary retention, increased body temperature, excessive sweating, pupil dilation, and sexual dysfunction.

Despite promising preliminary results from few initial studies, to date there have been no published replication studies or clinical trials of mirtazapine for treating ATS dependence in different populations and settings. The proposed study will provide additional data on tolerability, acceptability and potential efficacy of Mirtazapine for treatment of co-occurring opioid and ATS dependence (COATS) in Kelantan, Malaysia.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV criteria for both opioid and ATS dependence, as assessed by the Structured Clinical Interview for DSM (SCID)
2. Active COATS dependence as documented by ATS and opioid-positive urine tests and a report of at least 2 or more days per week of ATS use during the month prior to the study enrolment.
3. Age 18-65.

Exclusion Criteria:

1. Liver enzymes greater than 3 times the upper limit of normal or evidence of liver failure or acute hepatitis
2. Having serious medical or psychiatric illnesses (including current psychotic disorder, major depression, suicidal or homicidal ideations) or taking medications to treat depression or psychosis.
3. Refused informed consent or inability to understand the protocol or assessment questions

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of illicit ATS use. | 18 weeks
  This will be measured from baseline over time during treatment, based on urine toxicology testing and self-report

SECONDARY OUTCOMES:
Reductions in sexual and HIV risk behaviour iii) Improvement of social functioning | 18 weeks
  Measured by repeated assessments of sexual and HIV risk behaviours
Improvements in neuropsychological functioning | 18 weeks
  Measured by repeated assessments of neuropsychological functioning

CONTACTS AND LOCATIONS:
Overall Officials: Vicknasingam Kasinather, PhD, Principal Investigator — University Science Malaysia
Locations (1):
- University Science Malaysia, Kota Bharu, Kelantan, Malaysia